CLINICAL TRIAL: NCT07324616
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics of a Single Oral Dose of EDG-7500 in Participants With Impaired and Normal Hepatic Function
Brief Title: A Study to Evaluate EDG-7500 in Adults With Hepatic Impairment
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDG-7500-106
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Impairment (HI)
Keywords: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Adults (Experimental)
  Interventions: Drug: EDG-7500
- Mild Hepatic Impairment (Experimental)
  Interventions: Drug: EDG-7500
- Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: EDG-7500

INTERVENTIONS:
Drug: EDG-7500 — Single dose of EDG-7500

SUMMARY:
The purpose of this Phase 1 study is to understand and compare the amount of EDG-7500 in the blood after a single dose in participants with different levels of liver function impairment versus participants with normal liver function. The safety of EDG-7500 in adult participants with different levels of liver function impairment will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* Adult, male or female, ≥ 18 years of age.
* Female and male participants must follow protocol-specified contraception guidance.
* Continuous non-smoker or moderate smoker (≤ 10 cigarettes per day or equivalent) for at least 3 months prior to dosing.
* BMI ≥ 18.0 and ≤ 40.0 kg/m2 at screening.
* eGFR >60 mL/min calculated using the 2021 CKD-EPI creatinine equation.

Participants with Mild and Moderate Hepatic Impairment (HI)

* With the exception of HI, is in generally good health for study participation including the following:

  * Pulse rate is ≥ 40 bpm and ≤ 110 bpm at screening.
  * QTcF interval is ≤ 500 msec and has ECG findings considered normal or not clinically significant.
* Has impaired hepatic function as defined by the Child-Pugh classification for severity of liver disease and has a Child-Pugh score in line with one of the following HI cohorts at screening:

  * Mild HI (Class A): Child-Pugh score of 5 to 6, inclusive.
  * Moderate HI (Class B): Child-Pugh score of 7 to 9, inclusive.
* Has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency.

Participants with Normal Hepatic Function:

-Medically healthy, including the following:

* Blood pressure is ≥ 90/40 mmHg and ≤ 150/95 mmHg.
* Pulse rate is ≥ 40 bpm and ≤ 100 bpm.
* QTcF interval is ≤ 470 msec and has ECG findings considered normal or not clinically significant.
* Liver function test including ALT ≤ ULN, AST ≤ ULN, and total bilirubin ≤1.5x ULN.

Exclusion Criteria:

All Participants

* History or presence of alcohol or drug abuse within the past 1 year prior to dosing.
* Female participant with a positive pregnancy test at the screening visit or at check-in or who is lactating or breastfeeding.
* Positive urine or breath alcohol results at screening or check-in. Unable to refrain from or anticipates the use of any drugs.
* Positive results for HIV at screening.
* Donation of blood or significant blood loss within 56 days prior to dosing.
* Plasma donation within 7 days prior to dosing.
* Participation in another clinical study within 30 days or within 5 half-lives (if known), prior to dosing.

Participants with Mild and Moderate HI

* With the exception of HI, history or presence of clinically significant medical or psychiatric condition or disease, or any illness that might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* History of severe complications of liver disease within the preceding 3 months of screening.
* Primary biliary cholangitis or biliary obstruction at screening.
* Fluctuating or rapidly deteriorating hepatic function from screening until prior to dosing.
* History of liver or other solid organ transplantation.
* Requires paracentesis more often than 2 times per month.
* Transjugular intrahepatic portosystemic shunt and/or has undergone portacaval shunting within 90 days prior to screening.
* Received antiviral and/or immune modulating therapy for active hepatitis infection within 90 days prior to dosing.
* Diabetic participants with HbA1c > 8.5% at screening.
* Positive for HBsAg or HBcAb and has positive hepatitis B virus DNA at screening.
* Positive for HCV and has a detectable HCV viral load at screening.

Participants with Normal Hepatic Function

* History or presence of clinically significant medical or psychiatric condition or disease, or any illness that might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Alcohol consumption > 14 drinks per week for males (7 for females) within 45 days of screening.
* Positive result for HBsAg or HCV at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration time-curve from time zero to the last measured concentration (AUC0-last) | Pre-dose to day 10
Area under the plasma concentration time-curve from time zero extrapolated to infinity (AUC0-inf) | Pre-dose to day 10
Maximum observed plasma concentration (Cmax) | Pre-dose to day 10

SECONDARY OUTCOMES:
Safety: incidence of treatment-emergent adverse events | Up to 14 days of monitoring
  To evaluate the safety and tolerability of a single oral dose of EDG-7500 in participants with mild and moderate hepatic impairment and participants with normal hepatic function

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No